CLINICAL TRIAL: NCT00064740
Title: Relaxation Response With Acupuncture for HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001276-01A1 (NIH)
Record Dates: First submitted 2003-07-11; First posted 2003-07-14 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Human Immunodeficiency Virus; AIDS
Keywords: Human Immunodeficiency Viruses; Relaxation; Acupuncture; Complementary therapies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: relaxation response

SUMMARY:
Advances in treatment has turned HIV/AIDS into a chronic illness. Relaxation response is a state in which individuals evoke a bodily calm, effecting physiological changes that are shown to be associated with improved immune functioning. Acupuncture and relaxation are thought to both induce calm and deep relaxation in mind and body. This trial will study the combined effects of acupuncture and relaxation response in HIV patients.

DETAILED DESCRIPTION:
HIV/AIDS patients experience a range of symptoms associated with clinical manifestations of the disease, opportunistic infections, and medication side effects, all of which are strongly associated with quality of life (QoL). Many HIV/AIDS patients use complementary and alternative medicine (CAM) to help alleviate their symptoms and to improve their QoL. Among the various CAMs, acupuncture and relaxation response are commonly used regimens. These two therapies are thought to share common features and can complement each other in that acupuncture facilitates the effect of relaxation response and on the other hand relaxation response prepares the body to be more accessible to acupuncture. This study will test the feasibility of conducting a double blind 2-arm controlled trial and to collect pilot data in preparation for a large-scale study to fully test the hypothesis that adding relaxation response to acupuncture will have an enhanced effect in HIV+ patients. For this pilot study, we will recruit 100 HIV+ patients who are currently receiving acupuncture. Study participants in the intervention group will listen to tapes with instructions to elicit the relaxation response as well as music routinely played while receiving acupuncture. Study participants in the control group will receive usual care that is listening to music while receiving acupuncture. Study participants in the intervention group will be given the relaxation response tapes for home practice and they are asked to record the frequency of usage. We will assess both groups' symptoms and quality of life at baseline, 4 weeks, 8 weeks, and upon completion of the intervention at 12 weeks. We will assess the feasibility using various indicators, including patient evaluation of the study. Ultimately, the qualitative analysis of patients' study evaluation as well as the longitudinal regression analysis results that compare the outcomes between the intervention and control groups will be used to help design a future large-scale study of the relaxation response intervention among HIV+ patients treated with acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* First time and long-term acupuncture users
* Symptomatic criteria including: sinus problem, headache, dental pain/sore or bleeding gums, nausea, diarrhea, vomiting, muscle aches, joint pain, neuropathy, weakness, anxiety, depression, and insomnia

Exclusion Criteria:

* Patients suffering from acute symptoms
* Patients with acute opportunistic infections
* Patients currently practicing relaxation response
* Patients currently enrolled in another intervention study
* Cognitive impairment as measured by MMSE (Mini Mental Status Examination)
* Lack of English proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-07; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Bei-Hung Chang, Sc.D, Principal Investigator — Assistant Professor at Boston University School of Public Health
Locations (1):
- Aids Care Program, Boston, Massachusetts, United States